CLINICAL TRIAL: NCT05312203
Title: A Randomized Control Trial to Investigate the Effectiveness of Smart Mental Health Interventions for Stress Reduction(inMind) During the Pharmacological Treatment in Mild to Moderate Major Depressive Disorder.
Brief Title: Alleviating Stress by Mobile Application' for Depression
Acronym: ASMA-D
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korea University Guro Hospital (Other)
Collaborators: Ministry of Trade, Industry & Energy, Republic of Korea (Other Government)
Responsible Party: Principal Investigator, Han, Chang Su, Professor, Korea University Guro Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021GR0585
Record Dates: First submitted 2022-03-23; First posted 2022-04-05 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-11

CONDITIONS: Major Depressive Disorder
Keywords: Stress; Major depressive disorders; Mobile health; Mindfulness-based intervention; Cognitive-behavior therapy; Relaxation Therapy; Cost-effectiveness; Randomised controlled trial
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: This study is a single-blind, multicenter, randomized, controlled crossover trial.
Who Masked: Outcomes Assessor
Masking Description: Due to the intervention's nature, this will be a single-blind study in which the results will be assessed blindly, but participants will be aware of their group assignment. Most of the assessments are self-rated, and the clinician rating, HAM-D, will be assessed by an independent blinded evaluator not participating in the assignment and care providing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the App first group (fAPP) (Other): Participants assigned to fAPP group will use the App initially for 28 consecutive days (T1). After T1, during the next 28 consecutive days (T2) without washout period, fAPP will only maintain the usual treatment.
  Interventions: Other: the App
- wait list crossover group (dAPP) (Other): During T1, participants assigned to the dAPP arm will maintain the usual treatment. After T1, during the next 28 consecutive days (T2) without washout period, dAPP will use the APP.
  Interventions: Other: the App

INTERVENTIONS:
Other: the App — The App provides content for mobile-based stress relief that can be used on most Android and iOS-based mobile devices. Content for stress relief consists of three modules; meditation, cognitive approach, and relaxation sounds. Additionally, the App includes the module for objective stress monitoring. The APP was originally designed and developed in Korean, but English, Chinese, and Japanese versions are also available. For use in the treatment environment, the manufacturer also provides a service that allows therapists to check their patients' application usage and their stress level measured by the stress monitoring module.
  Other Names: Integrated mobile application for stress reduction; "inMind" (Demand, Republic of Korea, http://www.demand.co.kr)

SUMMARY:
This study is a single-blind, multicenter, randomized, controlled crossover trial. The App, developed in South Korea, is an application that provides integrated interventions for stress reduction for the general population. The App provides three contents based on MBSR, CBT, and relaxation sounds that are known to be effective in stress reduction ("Meditation category", "Cognitive approach", and "Relaxation Sound", respectively). Participants (n = 215) recruited via medical practitioner referral will be randomized to App first group (fAPP) or a waitlist crossover group (dAPP). Inclusion criteria are age 19-65; diagnosed with mild to moderate major depressive disorders (Score of 7-24 on the Hamilton Rating Scale for Depression); Stable medication for 28 days prior to study participation. The study was conducted over eight weeks, the fAPP group used The App for the first four weeks and the dAPP group for the next four weeks, and during all study periods, the participants received usual pharmacological treatment. Primary outcome measures are the Depression Anxiety Stress Scale-21. The analysis will use mixed-model repeated measures.

DETAILED DESCRIPTION:
This study is a single-blind, multicenter, randomized, controlled crossover trial. All subjects who met the inclusion and exclusion criteria will be randomly assigned to the App first group (fAPP) and or a waitlist crossover group (dAPP). Due to the intervention's nature, this will be a single-blind study in which the results will be assessed blindly but participants will be aware of their group assignment. Participants assigned to fAPP group will use the App initially for 28 consecutive days (T1). During T1, participants assigned to the dAPP arm will maintain the usual treatment. After T1, during the next 28 consecutive days (T2) without washout period, dAPP will use the APP, and fAPP will only maintain the usual treatment. We assumed that there would be no carry-over effect as the App utilized in this study is not a curative treatment but rather a tool for relieving stress in patients with depression. Therefore, we decided to use a cross-over design without a wash-out period.

The three University Hospitals in the Republic of Korea participating in the study will recruit depressive patients for applying the App. The Korea University Guro Hospital and Korea University Anam Hospital are in the inner center of the Capital, and Korea University Ansan Hospital is in Ansan city, outskirts of the capital area. Each hospital is a general hospital, and the Korea University Guro Hospital will lead the ASMA-D study as. For patient recruitment, 96 patients (48 interventions and 48 controls) in the Korea University Guro Hospital and 60 patients (30 interventions and 30 controls) in each from Korea University Anam Hospital and Korea University Ansan Hospital will be expected.

Screening will begin for those who are interested in advertisements posted in the participating hospital among the depressive patients who visit the hospital. After interested patients will contact the research team. the patients will be screened for eligibility according to the above-described criteria by the psychiatrist. After eligibility is confirmed, details of study will be explained to potential participant. Once participant agrees to participate, Informed consent is obtained, patient is enrolled, and randomization only occurs after enrollment.

Successful volunteers will be randomly assigned to the fAPP of dAPP. Randomization is conducted using block randomization by each clinical center. To prevent bias towards one treatment group, eight patients will be configured in blocks and will be randomly assigned to groups fAPP and dAPP within each block. For consistent allocation, randomization will be done using a pre-built program. This program is created by Korea University Guro Hospital to blind the researcher from the information of assignment in advance.

Assessments are obtained clinician rating scale and self-rating scales during hospital visits. Assessments conducted at the hospital visit were acquired at the baseline (V0) and every two weeks (V1, V2, V3, and V4) during T1 and T2. The baseline assessments will be collected when participants are enrolled and include sociodemographic and clinical characteristics. All instruments have been translated to Korean with reliable psychometric properties. The data collection process implanted in the evaluation module of the mobile App will be activated through an ID issued after enrollment and randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Adults between the ages of 19 and 65;
2. Diagnosed with mild to moderate major depressive disorders in an expert interview evaluation according to the DSM-IV diagnostic criteria (Score of 7-24 on the Hamilton Rating Scale for Depression [HAM-D]);
3. Stable medication for 28 days prior to study participation;
4. Informed consent and voluntary participation.

Exclusion Criteria:

1. Hard to use smart phone or unable to independently use Application;
2. Diagnosed with severe major depressive disorder in an expert interview evaluation according to the DSM-5 diagnostic criteria (score of 25 or more on HAM-D);
3. Severe mental disorders (current or in the past), including Major depressive disorder with psychotic features, bipolar affective disorder, personality disorder, obsessive compulsive disorder, autism spectrum disorder, substance use disorder;
4. History of brain injury, epileptic seizures, intellectual disability, or cognitive disorders;
5. History of severe physical disorders, including cancer, tuberculosis, severe cardiovascular disease, etc.
6. Individuals participating in other cognitive behavioral therapy or activities related to stress relief

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-05-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Depression, Anxiety and Stress Scale (DASS-21) | Baseline / 2 week / 4 week / 6 week / 8 week
  DASS-21 is s a self-report measure of anxiety, depression and stress levels used in diverse settings developed by Lovibond [47]. The Korean version of DASS-21 was developed by Eun-Hyun Lee in 2018 [48]. This version was tested in Korean speaking samples and indicated that the items had been adequately and appropriately translated and adapted. Korean version of DASS-21 was tested in 481 Korean adults, the result showed that the Cronbach's α was 0.93.

SECONDARY OUTCOMES:
Change in Perceived stress scale (PSS) | Baseline / 4 week / 8 week
  The perceived stress scale (PSS) is used to measure the extent to which respondents feel that their stress is unpredictable, uncontrollable and overwhelming (e.g. In the last month, how often have you felt you were unable to control the important things in your life?) [49]. The validated Korean short version of the perceived stress scale (K-PSS) was used in the present study [50]. The K-PSS is a 10-item self-report questionnaire using a five-point Likert scale ranging from 0 (never) to 4 (very often). Total scores range from 0 to 40, with higher scores indicative of greater perceived stress (Cronbach's α = 0.819).
Change in Posttraumatic embitterment disorders scale (PTED) | Baseline / 4 week / 8 week
  Post Traumatic Embitterment Disorder Self-Rating Scale (PTED Scale) is designed to assess the features of embitterment reactions to negative life events [51]. Consisting of 19 items, the PTED Scale asked participants to rate their reactions to each negative life event during recent years using a 5-point scale ranging from 0 (not true at all) to 4 (extremely true). A mean total score of 2.5 was used as a cut-off score to detect the clinically significant reactive embitterment [51]. The Korean version of the PTED Scale was translated and validated with good internal consistency (Cronbach's α = 0.962) [52].
Change in 9-item Patient Health Questionnaire (PHQ-9) | Baseline / 2 week / 4 week / 6 week / 8 week
  The 9-item version of the Patient Health Questionnaire (PHQ-9) was developed from the historical Primary Care Evaluation of Mental Disorders (PRIME-MD), which was shortened to maximize clinical usefulness [53]. This measure has been widely used in primary care settings for psychiatric purposes, with major depression diagnosed if 5 or more of the 9 symptoms have been present more than half the days of the past 2 weeks, one of these symptoms being either depressed mood or anhedonia. Each item is rated on a scale from 0 to 3, and the total score can range from 0 to 27. The total scores of ≥5, ≥10 and ≥15 represent mild, moderate and severe levels of depression severity [54]. The Korean version of the PHQ-9 was translated and validated with good internal consistency (Cronbach's α = 0.86) [55].
Change in Hamilton depression rating scale (HAM-D) | Baseline / 2 week / 4 week / 6 week / 8 week
  he Hamilton Depression Rating Scale (HAM-D) is an inventory of questions that is employed to detect and identify the intensity or severity of the signs and symptoms of depression in patients who have been diagnosed with clinical depression [56]. The 17-item version of the HAM-D is more commonly used than the 21-item version, which contains four additional items that measure symptoms related to depression, such as paranoia and obsession, rather than the severity of the depressive symptoms themselves. The Korean version of the HAM-D was translated and validated with good internal consistency (Cronbach's α = 0.76) [57].
Intervention engagement | 4 week for fAPP 8 week for dAPP
  Activities on the application such as number of visits, time in-between logins and number of usages of each category, will be assessed through track and change functionalities (log files). Data on how patients use online modules (frequency, duration, order, completion), how they rate them and to what extent they adhere, will also be obtained through usage statistics on the App online server. All patient information from the server will be encrypted via Hypertext Transfer Protocol Secure which ensures no external parties are able to view it during transfer. Data access from server is also authenticated by a passphrase which is supplied from the Study coordinator, ensuring only the research assistants will be able to request and review patient data.

CONTACTS AND LOCATIONS:
Overall Officials: Changsu Han, MD, PhD, Study Chair — Department of Psychiatry, Korea University Guro Hospital, Korea University College of Medicine; Junhyung Kim, MD, PhD, Principal Investigator — Department of Psychiatry, Korea University Guro Hospital, Korea University College of Medicine; Cheolmin Shin, MD, PhD, Principal Investigator — Department of Psychiatry, Korea University Ansan Hospital, Korea University College of Medicine; Kyu-Man Han, MD, PhD, Principal Investigator — Department of Psychiatry, Korea University Anam Hospital, Korea University College of Medicine
Locations (1):
- Department of Psychiatry, Korea University Guro Hospital, Seoul, Guro Gu, South Korea

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and analyzed during the current study will be available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: The time when all research processes have been completed and the relevant results are published.

REFERENCES:
- [Derived] Kim J, Shin C, Han KM, Lee MS, Jeong HG, Pae CU, Patkar AA, Masand PM, Han C. Investigating the effectiveness of a smart mental health intervention (inMind) for stress reduction during pharmacological treatment for mild to moderate major depressive disorders: Study protocol for a randomized control trial. Front Psychiatry. 2023 Mar 14;14:1034246. doi: 10.3389/fpsyt.2023.1034246. eCollection 2023. PMID 36998625